CLINICAL TRIAL: NCT04455165
Title: Factors Influencing Morbi-mortality in Right Anterior Minithoracotomy Approch for Aortic Valve Replacement Operated at Dijon University Hospital
Brief Title: Factors Influencing Morbi-mortality in Right Anterior Minithoracotomy Approch for Aortic Valve Replacement
Acronym: RVAOMITAVA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier La Chartreuse (Other)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, PI, Centre Hospitalier La Chartreuse
Other Study IDs: CCVT-RVAoMITAVARegistry
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RVAo MITAVA: Patient operated since 2009 for aortic valve replacement through right anterior minithoracotomy approch in Dijon Burgundy University Hospital
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — Aortic valve replacement with or without associated cardiac surgery (coronary bypass, mitral valve surgery,...)

SUMMARY:
Since 2009, positive experiences with right anterior minithoracotomy as an approach to aortic valve replacement are extensively practiced in our institution. The primary disease process for which patients are referred remains aortic stenosis. But more and more, we met older patients with both aortic stenosis and other cardiac pathology (coronary artery disease, other valvulopathy...). Even if minimally invasive valve surgery has been demonstrated to significantly improve postoperative course (reduced blood transfusion, pain, hospital lengths of stay) and to enhance postoperative recovery, when compared with a median sternotomy, it is however important to have medical data and statistics in order to better understand the factors influencing morbi-mortality and thereby to continue this improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 y-o who underwent aortic valve replacement

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient operated for aortic valve replacement with or without associated cardiac surgery from 2009 in Dijon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
30 days mortality incidence rates | 30 days
  Mortality from aortic valve replacement to 30 days post-surgery

SECONDARY OUTCOMES:
30 days morbidity incidence rates | 30 days
  Morbidity from aortic valve replacement to 30 days post-surgery (major adverse cardiac events)
Long-term morbimortality incidence rates | 10 years
  Morbimortality from aortic valve replacement up to 10 years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Catherine MORGANT, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- Cardiovascular and thoracic surgery Unit - Dijon University Hopital, Dijon, France

IPD SHARING:
Plan to Share IPD: No
All patients signed a institutional form prior to the procedure stating that they did not object to the use of their medical data for research purposes. Before inclusion, all patients (or a trusted person) were informed about the study and its objectives. No opposition was expressed.